CLINICAL TRIAL: NCT06386484
Title: Selective Head-and-neck Cooling on Biomarker Levels and Symptom Rating Following a Boxing Bout- Protocol for an Exploratory Randomized Trial
Brief Title: Selective Head-and-neck Cooling on Biomarker Levels and Symptom Rating Following a Boxing Bout
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019-05463
Record Dates: First submitted 2024-04-16; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Repetitive Head Impact; Selective Head and Neck Cooling

STUDY DESIGN:
Intervention Model Description: The PolarCap System consists of a high-powered portable cooling system, designed to reduce brain temperature by controlled cooling of the scalp and neck with a circulating coolant (PolarCap Coolant, PolarCool AB, Lund, Sweden). The coolant is maintained at 0°C and flows through a silicone-based head cap. An insulating neoprene cover is put on top of the cap for isolation.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Boxers (Experimental)
  Interventions: Device: PolarCap System
- Controls (No Intervention)

INTERVENTIONS:
Device: PolarCap System — The PolarCap Coolant flows through a silicone-based head cap. An insulating neoprene cover is put on top of the cap to isolate the cold. Using PolarCap system to selective head and neck cooling for 45 minutes post fight in boxing.
  Arms: Boxers

SUMMARY:
Young, healthy elite boxers ≥ 18 years old are recruited. Prior to, and immediately after a competitive boxing bout over 3x2 or 3x3 minutes, blood samples are drawn. Boxers are randomized to intervention or control management by 1:1 allocation prior to baseline testing. After the initial post-fight blood sample is drawn and symptom rating using the sports concussion assessment tool-5 (SCAT-5) has been collected, the boxers receive either acute selective head-and-neck cooling for 45 min, or routine post-fight management. The number of head impacts are counted in all boxers on match video recordings. In both groups, blood samples are drawn 45 minutes after the initial post-bout blood sample, as well as 3 and 6 days post-fight.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female elite boxers ≥18 years old
2. Cleared for participation by the medical staff of the Swedish Boxing Association.
3. Informed consent by each participant prior to the competitive event
4. No boxing fights or match sparring during the initial 6 days after their last boxing fight
5. Signed informed consent.

Exclusion Criteria:

1. >40 years old or <18 years old
2. Participation in competitive fights, match-sparring or any training causing additional head impacts during the first six post-fight days after being included in the study.
3. History of autoimmune neurological diseases or a neurodegenerative disorder.
4. History of previous traumatic brain injury resulting in an intracranial haemorrhage.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Selective head-and-neck cooling in boxing attenuates the release of brain injury biomarkers such as NFL and GFAP post fight. | 6 days
  NFL (Neurofilament light), GFAP (Glial fibrillary acidic protein)

SECONDARY OUTCOMES:
Selective head-and-neck cooling improves symptom rating post fight in boxing, using the Sports Concussion Assessment tool- 5 (SCAT-5). | 6 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Sciences Lund, Department of Neurosurgery, Sweden, Lund, Skåne County, Sweden

REFERENCES:
- [Derived] Al-Husseini A, Tegner Y, Blennow K, Zetterberg H, Marklund N. Effects of Selective Head-and-Neck Cooling on Brain Injury-Related Biomarker Levels and Symptom Rating Following a Boxing Bout: Protocol for an Exploratory Randomized Trial. JMIR Res Protoc. 2025 Jun 16;14:e68954. doi: 10.2196/68954. PMID 40523276